CLINICAL TRIAL: NCT02218606
Title: An Exploratory Randomized Phase II Multicenter Trial of Abiraterone Acetate With or Without Cabazitaxel in Treatment of Metastatic Castration Resistant Prostate Cancer
Brief Title: Multicenter Trial of Abiraterone Acetate With or Without Cabazitaxel in Treatment of Metastatic Castration Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Sanofi (Industry); Thomas Jefferson University (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-046; PCCTC LOI: c12-108
Record Dates: First submitted 2014-08-08; First posted 2014-08-18 (Estimated); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer
Keywords: Abiraterone Acetate; CABAZITAXEL; CASTRATION RESISTANT; 14-046; Prostate Cancer Clinical Trials Consortium
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; cabazitaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abiraterone acetate 1000 mg po daily + prednisone 5 mg po BID (Experimental): Arm 1: Abiraterone acetate 1000 mg po daily + prednisone 5 mg po BID
  Interventions: Drug: Abiraterone acetate 1000 mg po daily; Drug: prednisone 5 mg po BID
- Cabazitaxel 25 mg/m2 IV + abiraterone acetate 1000 mg po daily (Experimental): Arm 2: Cabazitaxel 25 mg/m2 IV + abiraterone acetate 1000 mg po daily + prednisone 5 mg po BID
  Interventions: Drug: Abiraterone acetate 1000 mg po daily; Drug: Cabazitaxel 25 mg/m2 IV; Drug: prednisone 5 mg po BID

INTERVENTIONS:
Drug: Abiraterone acetate 1000 mg po daily
Drug: Cabazitaxel 25 mg/m2 IV
  Arms: Cabazitaxel 25 mg/m2 IV + abiraterone acetate 1000 mg po daily
Drug: prednisone 5 mg po BID

SUMMARY:
The purpose of this study is to see what effects (good and bad) treatment with abiraterone acetate (an oral hormonal agent) and prednisone (a steroid) with and without cabazitaxel (a chemotherapy) have on the cancer and to find out more about whether specific laboratory tests on tumor are useful in predicting how the patient will respond to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient needs to have a histologic or cytologic diagnosis of prostate cancer

Documented progressive metastatic CRPC based on at least one of the following criteria:

1. PSA progression defined as 25% increase over baseline value with an increase in the absolute value of at least 2 ng/mL that is confirmed by another PSA level with a minimum of a 1 week interval and a minimum PSA of 2 ng/mL.
2. Soft-tissue progression defined as an increase ≥ 20% in the sum of the LD of all target lesions based on the smallest sum LD since treatment started or the appearance of one or more new lesions.
3. Progression of bone disease (evaluable disease) or (new bone lesion(s)) by bone scan.

   * Agree to undergo a biopsy of at least one metastatic site or primary prostate for determination of the RB status. Adequate archival metastatic tissue can be used if available in lieu of a biopsy if done when patient had CRPC (within 6 months of treatment start).
   * ECOG performance status of 0-2.
   * Age ≥ 18 years.
   * Have testosterone < 50 ng/dL. Patients must continue primary androgen deprivation with an LHRH/GnRH analogue (agonist or antagonist) if they have not undergone orchiectomy.
   * Patients on long term (>6 months) anti-androgen therapy (e.g. flutamide, bicalutamide, nilutamide) will need to be off anti-androgen for 4 weeks (wash out period) and show evidence of disease progression off the anti-androgen. Patients that have been on an anti-androgen 6 months or less will need to discontinue anti-androgen therapy prior to treatment start (no wash out period required).
   * Patients must have adequate organ and marrow function as defined below obtained within 14 days prior to treatment start:
   * ANC >=1,500/μl
   * Hemoglobin >=9g/dL
   * Platelet count >=100,000/μl
   * Creatinine ≤ 1.5 x the institutional upper limit of normal (ULN)
   * Potassium > 3.5 mmol/L (within institutional normal range)
   * Bilirubin ≤ ULN (unless documented Gilbert's disease)
   * SGOT (AST) <=2.5 x ULN
   * SGPT (ALT) <=2.5 x ULN
   * The effects of cabazitaxel and abiraterone acetate on the developing human fetus at the recommended therapeutic dose are unknown. Men must agree to use adequate contraception prior to study entry, for the duration of study participation and for at least 3 months thereafter.
   * Patients must be able to take oral medication without crushing, dissolving or chewing tablets.
   * Patients may have received prior radiation therapy or major surgery. However, at least 21 days prior to treatment start must have elapsed since completion of radiation therapy or major surgery and patient must have recovered from all side effects at the time of randomization.
   * Ability to understand and the willingness to sign a written informed consent document that is approved by the local institutional review board.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents. Any prior investigational therapeutic products must be stopped at least 28 days (4 week washout) prior to treatment start.
* No prior exposure to abiraterone acetate or other specific CYP-17 inhibitors.
* No prior chemotherapy regimen. Prior isotope therapy with Strontium-89, Samarium or RAD223 should be completed at least three months (12 weeks) prior to treatment start.
* No ≥ grade 2 peripheral neuropathy
* Patients who have had antifungal agents (itraconazole, fluconazole) within 4 weeks prior to treatment start or those who have not recovered from AEs due to these agents administered more than 4 weeks earlier.
* Patients with a history of pituitary or adrenal dysfunction, active or symptomatic viral hepatitis or chronic liver disease are not eligible.
* Patients with known symptomatic brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other AEs.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cabazitaxel or other drugs formulated with polysorbate 80; or abiraterone acetate.
* Patients may continue on a daily Multi-Vitamin, calcium and Vitamin D, but all other herbal, alternative and food supplements (i.e. PC-Spes, Saw Palmetto, St John Wort, etc.) must be discontinued before treatment start. Patients must not be planning to receive any concurrent cytotoxic chemotherapy, surgery for their prostate cancer, or radiation therapy during protocol treatment.
* Patients on stable doses of bisphosphonates or the RANK-L inhibitor, Denosumab, which have been started no less than 4 weeks prior to treatment start, may continue on this medication, however patients are not allowed to initiate bisphosphonate/Denosumab therapy during the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III and IV heart failure), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Slovin, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Virginia Oncology Associates, Norfolk, Virginia

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Abiraterone Acetate 1000 mg po Daily + Prednisone 5 mg po BID: Arm 1: Abiraterone acetate 1000 mg po daily + prednisone 5 mg po BID
  Abiraterone acetate 1000 mg po daily
  prednisone 5 mg po BID
- Cabazitaxel 25 mg/m2 IV + Abiraterone Acetate 1000 mg po Daily: Arm 2: Cabazitaxel 25 mg/m2 IV + abiraterone acetate 1000 mg po daily + prednisone 5 mg po BID
  Abiraterone acetate 1000 mg po daily
  Cabazitaxel 25 mg/m2 IV
  prednisone 5 mg po BID
Period: Overall Study
Arm/Group | Abiraterone Acetate 1000 mg po Daily + Prednisone 5 mg po BID | Cabazitaxel 25 mg/m2 IV + Abiraterone Acetate 1000 mg po Daily
Started | 42 | 39
Completed | 17 | 7
Not Completed | 25 | 32
Not completed — Adverse Event | 1 | 1
Not completed — Death | 15 | 28
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Noncompliance | 1 | 0
Not completed — Initiation of new drug for prostate cancer | 2 | 0
Not completed — Other | 2 | 1
Not completed — Never started treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abiraterone Acetate 1000 mg po Daily + Prednisone 5 mg po BID | Cabazitaxel 25 mg/m2 IV + Abiraterone Acetate 1000 mg po Daily | Total
Number analyzed (Participants) | 42 | 39 | 81
Age, Continuous [Median (Full Range); unit: years] | 69.5 [50 to 85] | 67 [49 to 81] | 67 [49 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 42 | 39 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 42 | 39 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 34 | 29 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 39 | 81

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (rPFS)
Description: using the RECIST criteria
Time Frame: Up to 100 weeks
Measure: Median (Full Range); unit: months
Arm/Group | Abiraterone Acetate 1000 mg po Daily + Prednisone 5 mg po BID | Cabazitaxel 25 mg/m2 IV + Abiraterone Acetate 1000 mg po Daily
Number analyzed (Participants) | 42 | 39
months | 6.4 [3.8 to 10.6] | 14.8 [10.6 to 16.4]

2. Secondary Outcome: PSA Progression Free Survival (PSA PFS)
Description: For each patient, use a waterfall plot to report the percent change in PSA from baseline to 12 weeks (or earlier for those who discontinue therapy) and the maximum decline in PSA that occurs at any point after treatment.
Time Frame: Up to 100 weeks
Measure: Median (Full Range); unit: months
Arm/Group | Abiraterone Acetate 1000 mg po Daily + Prednisone 5 mg po BID | Cabazitaxel 25 mg/m2 IV + Abiraterone Acetate 1000 mg po Daily
Number analyzed (Participants) | 42 | 39
months | 9.2 [7.4 to 13.4] | 15.1 [10.9 to 19]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: per RECIST criteria
Time Frame: 1 year
Population: N/A - data were not collected
Arm/Group | Abiraterone Acetate 1000 mg po Daily + Prednisone 5 mg po BID | Cabazitaxel 25 mg/m2 IV + Abiraterone Acetate 1000 mg po Daily
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Participants With Maximum Overall Grade ≥3 AEs
Description: The NCI CTCAE version 4.0 will be used for recording and grading AEs.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone Acetate 1000 mg po Daily + Prednisone 5 mg po BID | Cabazitaxel 25 mg/m2 IV + Abiraterone Acetate 1000 mg po Daily
Number analyzed (Participants) | 42 | 39
Participants
  Participants with maximum overall grade ≥3 AEs | 27 | 23
  Participants without maximum overall grade ≥3 | 15 | 16

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Abiraterone Acetate 1000 mg po Daily + Prednisone 5 mg po BID | Cabazitaxel 25 mg/m2 IV + Abiraterone Acetate 1000 mg po Daily
All-Cause Mortality (participants affected / at risk) | 15/42 | 28/39
Serious Adverse Events (participants affected / at risk) | 22/42 | 28/39
Other Adverse Events (participants affected / at risk) | 27/42 | 23/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate 1000 mg po Daily + Prednisone 5 mg po BID (N=42) | Cabazitaxel 25 mg/m2 IV + Abiraterone Acetate 1000 mg po Daily (N=39)
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Acute kidney injury (Renal and urinary disorders) | 2 | 2
Anemia (Blood and lymphatic system disorders) | 1 | 4
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Creatinine increased (Investigations) | 1 | 0
Death NOS (General disorders) | 15 | 28
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Esophageal hemorrhage (Gastrointestinal disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Fatigue (General disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 4
Fever (General disorders) | 2 | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Hematoma (Vascular disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 2 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Lung infection (Infections and infestations) | 2 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Neutrophil count decreased (Investigations) | 2 | 2
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 6 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 2 | 1
Serum amylase increased (Investigations) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 1 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate 1000 mg po Daily + Prednisone 5 mg po BID (N=42) | Cabazitaxel 25 mg/m2 IV + Abiraterone Acetate 1000 mg po Daily (N=39)
Abdominal pain (Gastrointestinal disorders) | 8 | 6
Agitation (Psychiatric disorders) | 2 | 0
Alanine aminotransferase increased (Investigations) | 3 | 2
Alkaline phosphatase increased (Investigations) | 4 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3
Anemia (Blood and lymphatic system disorders) | 4 | 3
Anorexia (Metabolism and nutrition disorders) | 12 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 10
Blurred vision (Eye disorders) | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Bronchial infection (Infections and infestations) | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 4 | 1
Constipation (Gastrointestinal disorders) | 16 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 14
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Depression (Psychiatric disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 14 | 13
Dizziness (Nervous system disorders) | 4 | 5
Dry Mouth (Gastrointestinal disorders) | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 3
Dysgeusia (Nervous system disorders) | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 | 13
Edema limbs (General disorders) | 10 | 5
Fall (Injury, poisoning and procedural complications) | 3 | 0
Fatigue (General disorders) | 27 | 23
Fever (General disorders) | 3 | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Gait disturbance (General disorders) | 5 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 3
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Headache (Nervous system disorders) | 6 | 7
Hematuria (Renal and urinary disorders) | 8 | 8
Hot flashes (Vascular disorders) | 8 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 2
Hypertension (Vascular disorders) | 11 | 11
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Infection (Infections and infestations) | 3 | 1
Infections and infestations - Other, specify (Infections and infestations) | 3 | 2
Insomnia (Psychiatric disorders) | 0 | 6
Mucositis (Gastrointestinal disorders) | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 1 | 3
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 19 | 16
Nervous system disorders - Other, specify (Nervous system disorders) | 2 | 1
Neutrophil count decreased (Investigations) | 3 | 5
Non-cardiac chest pain (General disorders) | 2 | 1
Pain (General disorders) | 25 | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 7
Paresthesia (Nervous system disorders) | 1 | 2
Pelvic Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Peripheral Edema (General disorders) | 2 | 2
Peripheral motor neuropathy (Nervous system disorders) | 3 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 5
Platelet count decreased (Investigations) | 4 | 2
Pneumonia (Infections and infestations) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 2
Sensory Neuropathy (Nervous system disorders) | 0 | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 3
Upper respiratory infection (Infections and infestations) | 0 | 3
Urinary frequency (Renal and urinary disorders) | 16 | 17
Urinary incontinence (Renal and urinary disorders) | 9 | 13
Urinary retention (Renal and urinary disorders) | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 2
Urinary tract pain (Renal and urinary disorders) | 2 | 4
Urinary urgency (Renal and urinary disorders) | 5 | 4
Vomiting (Gastrointestinal disorders) | 7 | 11
Weight gain (Investigations) | 4 | 6
Weight loss (Investigations) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/06/NCT02218606/Prot_SAP_000.pdf